CLINICAL TRIAL: NCT05944718
Title: Three-arm Pragmatic Randomized Study on the Effectiveness, Feasibility, Acceptability, and Cost of the Use of Continuous Glucose Monitoring Devices Among People Living With Type 1 Diabetes in South Africa
Brief Title: Use of Continuous Glucose Monitoring Devices Among People Living With Type 1 Diabetes in South Africa
Acronym: ACCEDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); University of Pretoria (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NC008
Record Dates: First submitted 2023-06-19; First posted 2023-07-13 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
Keywords: continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Three arm pragmatic randomized controlled study Arm 1: use of CGM in a continuous manner from enrolment to the end of intervention period Arm 2: intermittent use of CGM (use for 2 weeks once every three months) from enrolment to the end of intervention period Arm 3 (control): standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): Arm 1 is those participants randomized to use of CGM in a continuous fashion; CGM use for the duration of 9 months.
  Interventions: Device: Continuous glucose monitor
- Arm 2 (Experimental): Arm 2 is those participants randomized to intermittent use of CGM; CGM use for 4 time points consisting of 2 weeks of CGM use each, for the duration of 9 months.
  Interventions: Device: Continuous glucose monitor
- Arm 3 (No Intervention): Arm 3 is those participants randomized to standard of care; regular use of self-monitoring of blood glucose (SMBG) for the duration of 9 months.

INTERVENTIONS:
Device: Continuous glucose monitor — Continuous Glucose Monitoring (CGM) is a technology used to measure glucose levels in people with diabetes. Unlike traditional finger prick self-monitoring of blood glucose (SMBG), CGM devices provide continuous and real-time glucose readings throughout the day and night.
  CGM systems consist of a small sensor that is inserted under the skin to measure glucose levels in the interstitial fluid, a transmitter that sends the glucose data to a receiver or smartphone, which shows the glucose readings. The sensor measures glucose levels automatically at regular intervals, eliminating the need for frequent finger pricks.
  CGM devices can track glucose trends, identify high or low glucose levels, and provide alerts for hypo- or hyperglycemia. This can help individuals make more informed decisions regarding their diabetes management, such as adjusting insulin doses, dietary choices, or physical activity levels.
  Other Names: Freestyle Libre Abbott
  Arms: Arm 1; Arm 2

SUMMARY:
Diabetes mellitus (diabetes) is a chronic condition that represents a major public health and clinical concern. Self-monitoring of blood glucose (SMBG) is a critical part of the care of individuals with diabetes. SMBG entails capillary fingerstick blood glucose testing multiple times per day. Many people with diabetes find this testing painful and cumbersome, often resulting in poor compliance to a glucose self-monitoring schedule. Furthermore, SMBG only provides limited visibility on daily and nightly glucose profiles, meaning that hypo- and hyperglycaemic episodes can be missed or detected with delay. The use of minimally invasive continuous glucose monitoring devices (CGMs) in diabetes management circumvents these challenges as CGMs measure glucose every few minutes over a period of 1-2 weeks through a sensor with a fine needle that is inserted once into a user's arm or abdomen. This enables periodic glucose measurement without repeat finger pricks and provides the user with a detailed glucose profile over the entire wear time of the sensor, thus enabling better adjustment of therapy or behaviour.

In populations where CGMs are accessible to people with diabetes as standard of care and without additional cost, many people with type 1 diabetes have switched from SMBG via fingerstick to the use of CGMs permanently, using the devices continuously. This is rarely possibly for people with type 1 diabetes in the public sector in LMICs as CGMs are not provided as standard of care. Little data on effectiveness, feasibility, acceptability, and cost of the use of CGMs in LMIC populations is available to inform clinical models for the integration of CGMs into diabetes management. Furthermore, it has not been investigated if intermittent, as opposed to continuous use of CGMs provides clinical benefit. Intermittent use could be beneficial for people with diabetes who do not have the means to pay for continuous use of CGMs.

This study aims to evaluate the effectiveness, feasibility, acceptability, and cost of intermittent and continuous use of CGM among people with type 1 diabetes in South Africa.

DETAILED DESCRIPTION:
3 Study Design As this study is a PrCT the study aspects will be embedded in the normal clinical care delivery of diabetes care in the selected clinics (see section 3.2, Scientific Rational for Selection of Study Design). Introducing only 1 additional clinic visit and 1 additional qualitative visit for study related procedures. The primary outcome measure, HbA1c, will be assessed through the HbA1c testing that is already used in these clinics. It is important to note that the type of HbA1c test (i.e.: laboratory-based vs point-of-care) per participant must remain constant during the study, this is because of variability of performance between various HbA1c testing platforms.

3.1 General Design This is a three-arm pragmatic randomized control study. The expected duration of study participants involvement in the study is 15 months, this consists of 9 months of intervention with a follow up visit 6 months post the last interventional study visit. There will be 6 total study visits for all participants.

* Arm 1 is those participants randomized to use of CGM in a continuous fashion; CGM use for the duration of 9 months.
* Arm 2 is those participants randomized to intermittent use of CGM; CGM use for 4 time points consisting of 2 weeks of CGM use each, for the duration of 9 months.
* Arm 3 is those participants randomized to standard of care; regular use of self-monitoring of blood glucose (SMBG) for the duration of 9 months.

For all participants the first study visit will consist of:

1. Enrolment including ICF,
2. Baseline surveys including demographics, the Glucose Monitoring Satisfaction Survey (GMSS-T1D), HRQOL surveys, and diabetes distress score survey.
3. Randomized assignment to study arm,
4. Blood draw for HbA1c testing (if not already done in the previous 1 month).

Those participants randomized to Arm 1 and Arm 2 will receive an education session on the CGM, be provided with the CGM, and be guided how to self-apply the CGM during enrolment visit.

During all Study Follow Up visits participants will have blood drawn for HbA1c testing, complete a brief survey to capture any hospitalizations and/or hypoglycaemic events related to diabetes complications that occurred between study visits.

Additionally, during Study Follow up visit C participants will complete the Glucose Monitoring Satisfaction Survey (GMSS-T1D), diabetes distress score survey, and an acceptability survey. During Study Follow up visit D, participants will complete the HRQOL surveys and diabetes distress score survey. During Study Follow up visit E participants will complete the Glucose Monitoring Satisfaction Survey (GMSS-T1D), diabetes distress score survey, and HRQOL surveys.

Detailed explanation of the study visits per arm are outlined below by arm in section 3.1.1, 3.1.2, 3.1.3

Qualitative methods used across all arms will consist of focus group discussions (FGDs) among the participants and caregivers of participants. Approximately 15 participants above the age of 18 years old will be selected from each arm (n=45, 3 FGD in total) and approximately 15 participants age range of 11 to 17 years old will be selected from each arm (n=45, 3 FGD in total) to participate in arm specific FGD to take place 30 to 35 weeks after study enrolment started. These FGDs will focus on understanding participant perceptions towards their current glucose monitoring devices and quality of life. To capture the perspectives of care givers of children and adolescents living with T1 diabetes 15 caregivers will be selected from each arm (n=45, 3 FGD in total) to participate in arm specific FGDs to take place 30 to 35 weeks after study enrolment started. These FGDs will focus on understanding care giver perspectives towards their minor's glucose monitoring devices and quality of life from the perspective of the care giver as well as their perceptions towards the quality of life for their minor.

Qualitative methods will also be used to gather perceptions from the healthcare providers regarding their perceptions surrounding the feasibility and acceptability of use of CGMs in their settings. This will consist of a semi-structured interviews (SSI) of selected HCW (n=10 total) to be conducted after week 36 after study enrolment started.

3.1.1 Arm 1 Continuous use of CGM For those in Arm 1 there will be 6 study visits for all participants. There will be an additional visit for a FGD among a subset of participants.

1. Enrolment visit: For those randomized to Arm 1 they will receive an education session on the CGM, be provided with the CGM, blood will be drawn for HbA1c testing (where this is standard of care) and be guided how to self-apply the CGM during enrolment visit.
2. Study Follow up A: The second study visit will take place 1 week after the enrolment visit. During this second visit the participant will see the clinician and review the CGM data from the first week. Participants in Arm 1 will be provided with 6 additional CGMs to continually use the CGM devices until their third study visit (Study Follow up B) to take place 12 weeks after enrolment.
3. Study Follow up B: At the third study visit participants will see the clinician and review the CGM data from the period of time in between second study visit and current, blood will be drawn for HbA1c testing, and the participant will be provided with 6 additional CGMS such that they continually use the CGM devices until their fourth study visit (Study Follow up C) to take place at 24 weeks after enrolment.
4. Study Follow up C: At the fourth study visit participants will see the clinician and review the CGM data from the period of time in between third study visit and current, blood will be drawn for HbA1c testing, and the participant will be provided with 6 additional CGMS such that the continually use the CGM devices until their fifth study visit (Study Follow up D) to take place at 36 weeks after enrolment.
5. Study Follow up D: At the fifth study visit participants will see the clinician and review the CGM data from the period in between fourth study visit and current, blood will be drawn for HbA1c testing and the participant will be provided with 1 additional CGM to use for the week following Study follow up C.
6. Study Follow up E: At the sixth and final study visit which takes place at 58 weeks after enrolment study participants will see the clinician and blood will be drawn for HbA1c.

3.1.2 Arm 2 Intermittent use of CGM For those in Arm 2 there will be 6 study visits for all participants. There will be an additional visit for a FGD among a subset of participants.

1. Enrolment visit: For those randomized to Arm 2 they will receive an education session on the CGM, be provided with the CGM, blood will be drawn for HbA1c testing, and be guided how to self-apply the CGM during enrolment visit.
2. Study Follow up A: The second study visit will take place 1 week after the enrolment visit. During this second visit the participant will see the clinician and review the CGM data from the first week. During Study follow up A participants in Arm 2 will be provided 1 CGM to use starting 1 week before their third study visit (Study Follow up B) to take place at 12 weeks after enrolment.
3. Study Follow up B: At the third study visit participants will see the clinician and review the CGM data from the preceding week before Study follow up A, blood will be drawn for HbA1c testing, and the participant will be provided with 1 additional CGM such that the participant uses the CGM for the week directly following Study follow up A and 1 week before their fourth study visit (Study Follow up C) to take place at 24 weeks after enrolment.
4. Study Follow up C: At the fourth study visit participants will see the clinician and review the CGM data from the preceding week before Study follow up B, blood will be drawn for HbA1c testing, and the participant will be provided with 1 additional CGM such that the participant uses the CGM for the week directly following Study follow up A, and 1 week before their fifth study visit (Study Follow up D) to take place 36 weeks after enrolment.
5. Study Follow up D: At the fifth study visit participants will see the clinician and review the CGM data from the week preceding Study Follow up D, blood will be drawn for HbA1c testing and the participant will be provided with 1 additional CGM to use for the week following Study follow up D.
6. Study Follow up E: At the sixth and final study visit which takes place at 58 weeks after enrolment study participants will see the clinicals and blood will be drawn for HbA1c.

3.1.3 Arm 3 Standard of Care For those in Arm 3 there will be 6 study visits for all participants. There will be an additional visit for a FGD among a subset of participants. Participants will follow the standard of care at each clinic.

1. Enrolment visit: Those participants randomized to Arm 3 will undergo blood drawn for HbA1c testing.
2. Study Follow up A: The second visit will take place 1 week after the enrolment visit. Participants will see their clinician at the enrolment visit as per SoC
3. Study Follow up B: The third study visit will take place at 12 weeks after enrolment, participants will see the clinician as per SoC. Blood will be drawn for HbA1c testing.
4. Study Follow up C: The fourth study visit will take place at 24 weeks after enrolment. participants will see the clinician as per SoC. Blood will be drawn for HbA1c testing.
5. Study Follow up D: The fifth study visit will take place at the end of 35 weeks after enrolment. Participants will see the clinician as per SoC. Blood will be drawn for HbA1c.
6. Study Follow up E: The sixth and final study visit will take place at 58 weeks after enrolment. participants will see the clinician as per SoC. Blood will be drawn for HbA1c. After completion of study participation, those in Arm 3 will be offered 1 CGM to use such that they can experience CGM use. Those participants who accept the CGM will be provided with an education session on CGM use before application.

3.2 Scientific Rationale for Study Design As this study intendeds to generate evidence to inform policy and decision makers on the potential benefits of use of CGM in South Africa a pragmatic, rather than an explanatory, randomized control study design was selected [9]. A PrCT design was selected as the study aims to understand the impact of CGM use in as close to real world settings as possible. A classically designed randomized control trial with overly strict study criteria and processes may lead results that are not directly translatable to real world experience, while a classical RCT may have strong internal validity often RCTs are criticized for a lack of external validity, therefore a PrCT design was selected to balance internal and external validity [12]. A PrCT design may "provide more realistic effect size estimates and enhance translation of research findings into clinical practice".

ELIGIBILITY:
Inclusion Criteria:

* Recipient of care participants are eligible to be included in the Study only if all the following inclusion criteria apply:

People living with T1 diabetes with HbA1c current levels ≥10% within the last 3 months (and at least 2 HbA1c ≥10% within the last 18 months prior to study enrolment) who are attending for diabetes care at the 3 study clinics.

* Care givers to children/adolescents living with T1 diabetes are eligible to be included in the study only if all the following inclusion criteria apply:

  • The child/adolescent that the person is a care giver to is enrolled in the study.
* Healthcare providers are eligible to be included in the study only if all the following inclusion criteria apply:

  * Healthcare provider at the study sties engaged in diabetes care provision related to the study.

Exclusion Criteria:

* Participants are excluded from the Study if any of the following exclusion criteria apply:

  * People living with T1 diabetes under 4 years old as this the minimum age for use of CGM as per the CGMs used in this study manufacturer instructions.
  * People diagnosed with T1 diabetes within the last 2 years.
  * People who have used a CGM in the last 6 months prior to enrollment.
  * People who anticipate that they would have access to a CGM through means outside this study during the duration of the study (15 months).
  * People living with Type 2 diabetes.
  * Known pregnancy at the time of study enrolment.
  * People who are not willing to agree to Freestyle Libre T&Cs

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Impact of continuous and intermittent CGM use on blood glucose levels in comparison to standard of care in people living with type 1 diabetes | 15 months
  Comparison of the magnitude of change in HbA1c levels before and after treatment in standard of care, continuous, and intermittent CGM arms

SECONDARY OUTCOMES:
1a. Impact of continuous and intermittent CGM use on the variability of blood glucose concentrations related to diabetes. | 15 months
  Estimates of coefficient of variation (CV) for glucose concentrations with 95% confidence intervals, for participants who received the CGM treatments.
1b. Impact of continuous and intermittent CGM use on the variability of blood glucose concentrations related to diabetes. | 15 months
  Estimates Time in Range (TIR) with 95% confidence intervals for participants who received the CGM treatments.
1c.Impact of continuous and intermittent CGM use on the variability of blood glucose concentrations related to diabetes. | 15 months
  Estimates Time Below Range (TBR) with 95% confidence intervals for participants who received the CGM treatments.
1d. Impact of continuous and intermittent CGM use on the variability of blood glucose concentrations related to diabetes. | 15 months
  Estimates Time Above Range (TAR) with 95% confidence intervals for participants who received the CGM treatments.
2. Impact of continuous and intermittent CGM use on unplanned visits to outpatient clinics and/or hospital related to diabetes complications. | 15 months
  Number of hospitalizations related to diabetes complications per each group, represented by means and standard deviations.
3a. Impact of continuous and intermittent CGM use on quality of life of recipients of diabetes care and their caregivers (where applicable) | 15 months
  Mixed methods QoL A: survey results including EQ-5D-Y/EQ-5D and Diabetes distress scores at baseline, midpoint, end point of intervention and endpoint of study.
3b. Impact of continuous and intermittent CGM use on quality of life of recipients of diabetes care and their caregivers (where applicable) | 15 months
  Mixed methods : Qualitative methods FGD among recipients of care and their caregivers
4a. Acceptability and feasibility of continuous and intermittent CGM use from a healthcare provider, recipients of care and care givers perspective. | 15 months
  Mixed methods: Feasibility will be assessed based on Arm 1 and Arm 2 adherence to protocol in terms of CGM use.
4b.Acceptability and feasibility of continuous and intermittent CGM use from a healthcare provider, recipients of care and care givers perspective. | 15 months
  survey from baseline, midline, and endline among recipients of care and their caregivers.
4c. Acceptability and feasibility of continuous and intermittent CGM use from a healthcare provider, recipients of care and care givers perspective. | 15 months
  Mixed methods: Qualitative methods: SSI among health care providers involved in clinical care at the study sites.
5. Cost of continuous and intermittent CGM use from a user and provider perspective | 15 months
  Costing surveys which capture direct and indirect costs at each follow-up visit among recipients of care, their caregivers and healthcare provider, and at end point of study, modelling over time horizon may be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Vetter, Study Director — Find
Locations (3):
- South Africa (3):
  - Steve Biko Academic Hospital, Pretoria, Gauteng
  - Groote Schuur Hospital - Diabetes Centre, Cape Town, Western Cape
  - Red Cross Hospital, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maiorino MI, Signoriello S, Maio A, Chiodini P, Bellastella G, Scappaticcio L, Longo M, Giugliano D, Esposito K. Effects of Continuous Glucose Monitoring on Metrics of Glycemic Control in Diabetes: A Systematic Review With Meta-analysis of Randomized Controlled Trials. Diabetes Care. 2020 May;43(5):1146-1156. doi: 10.2337/dc19-1459. PMID 32312858
- [Background] Lind M, Polonsky W, Hirsch IB, Heise T, Bolinder J, Dahlqvist S, Schwarz E, Olafsdottir AF, Frid A, Wedel H, Ahlen E, Nystrom T, Hellman J. Continuous Glucose Monitoring vs Conventional Therapy for Glycemic Control in Adults With Type 1 Diabetes Treated With Multiple Daily Insulin Injections: The GOLD Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):379-387. doi: 10.1001/jama.2016.19976. PMID 28118454
- [Background] Beck RW, Riddlesworth T, Ruedy K, Ahmann A, Bergenstal R, Haller S, Kollman C, Kruger D, McGill JB, Polonsky W, Toschi E, Wolpert H, Price D; DIAMOND Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Adults With Type 1 Diabetes Using Insulin Injections: The DIAMOND Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):371-378. doi: 10.1001/jama.2016.19975. PMID 28118453
- [Background] Welsh JB, Gao P, Derdzinski M, Puhr S, Johnson TK, Walker TC, Graham C. Accuracy, Utilization, and Effectiveness Comparisons of Different Continuous Glucose Monitoring Systems. Diabetes Technol Ther. 2019 Mar;21(3):128-132. doi: 10.1089/dia.2018.0374. Epub 2019 Jan 25. PMID 30681379
- [Background] Brown JVE, Ajjan R, Siddiqi N, Coventry PA. Acceptability and feasibility of continuous glucose monitoring in people with diabetes: protocol for a mixed-methods systematic review of quantitative and qualitative evidence. Syst Rev. 2022 Dec 9;11(1):263. doi: 10.1186/s13643-022-02126-9. PMID 36494845
- [Background] Distiller LA, Cranston I, Mazze R. First Clinical Experience with Retrospective Flash Glucose Monitoring (FGM) Analysis in South Africa: Characterizing Glycemic Control with Ambulatory Glucose Profile. J Diabetes Sci Technol. 2016 Nov 1;10(6):1294-1302. doi: 10.1177/1932296816648165. Print 2016 Nov. PMID 27154973
- [Background] Wells, R. and Knowles, A., 2023. The psychological and health benefits of using a continuous glucose monitor for a person with type 1 diabetes: A South African higher education context. F1000Research, 12(373), p.373.
- [Background] van Heerden, A., Kolozali, Ş. and Norris, S.A., 2022. Feasibility and acceptability of continuous at-home glucose monitoring during pregnancy: a mixed-methods pilot study. South African Journal of Clinical Nutrition, pp.1-8.
- [Background] Gamerman, V., Cai, T. and Elsäßer, A., 2019. Pragmatic randomized clinical trials: best practices and statistical guidance. Health Services and Outcomes Research Methodology, 19, pp.23-35.
- [Background] Treweek S, Zwarenstein M. Making trials matter: pragmatic and explanatory trials and the problem of applicability. Trials. 2009 Jun 3;10:37. doi: 10.1186/1745-6215-10-37. PMID 19493350
- [Background] Hohenschurz-Schmidt DJ, Cherkin D, Rice ASC, Dworkin RH, Turk DC, McDermott MP, Bair MJ, DeBar LL, Edwards RR, Farrar JT, Kerns RD, Markman JD, Rowbotham MC, Sherman KJ, Wasan AD, Cowan P, Desjardins P, Ferguson M, Freeman R, Gewandter JS, Gilron I, Grol-Prokopczyk H, Hertz SH, Iyengar S, Kamp C, Karp BI, Kleykamp BA, Loeser JD, Mackey S, Malamut R, McNicol E, Patel KV, Sandbrink F, Schmader K, Simon L, Steiner DJ, Veasley C, Vollert J. Research objectives and general considerations for pragmatic clinical trials of pain treatments: IMMPACT statement. Pain. 2023 Jul 1;164(7):1457-1472. doi: 10.1097/j.pain.0000000000002888. Epub 2023 Mar 22. PMID 36943273
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Cohen, J., 1988. Statistical power analysis for the behavioral sciences (2nd ed.). Hillsdale, NJ: Erlbaum.
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Bowen, G.A., 2008. Naturalistic inquiry and the saturation concept: a research note. Qualitative research, 8(1), pp.137-152.
- [Derived] Marban-Castro E, Muhwava L, Kamau Y, Safary E, Rheeder P, Karsas M, Kemp T, Freitas J, Carrihill M, Dave J, Katambo D, Kimetto J, Allie R; Kenya ACCEDE study group; South Africa ACCEDE study group; Ndungu J, Sigwebela N, Akach D, Girdwood S, Erkosar B, Nichols BE, Haldane C, Vetter B, Shilton S. Implementation research: a protocol for two three-arm pragmatic randomised controlled trials on continuous glucose monitoring devices in people with type 1 diabetes in South Africa and Kenya. Trials. 2024 May 21;25(1):331. doi: 10.1186/s13063-024-08132-7. PMID 38773658